CLINICAL TRIAL: NCT06366568
Title: Clinical Investigation to Assess the Efficacy of a Eugenol-based Product in Improving the Quality of Toothbrushing Measured by Plaque Assessment and Patient Perception Questionnaire and Relieving Gum Discomfort Areas
Brief Title: Efficacy of a Eugenol-based Product to Improve the Quality of Toothbrushing and Relieving Gum Discomfort Areas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRO-2022-10-PG-MER-MW-JG
Record Dates: First submitted 2024-04-03; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Plaque, Dental
Keywords: plaque gingivitis
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): toothpaste and gum product, brushing 2x a day for 2 minutes followed by gum product application
  Interventions: Drug: fluoride toothpaste containing 1450 ppm of MFP in a PCC base and eugenol gum product
- Group 2 (Placebo Comparator): toothpaste , brushing 2x a day for 2 minutes
  Interventions: Drug: fluoride toothpaste containing 1450 ppm of MFP in a PCC base

INTERVENTIONS:
Drug: fluoride toothpaste containing 1450 ppm of MFP in a PCC base and eugenol gum product — PARTICIPANTS WILL USE A EUGENOL BASED product PRIOR TO TOOTHBRUSHING
  Arms: Group 1
Drug: fluoride toothpaste containing 1450 ppm of MFP in a PCC base — toothbrushing 2x a day for 2 minutes each time
  Arms: Group 2

SUMMARY:
The objective of this study is to evaluate the efficacy of a eugenol-based product in improving the quality of toothbrushing and relieving areas of gingival discomfort. This is a randomized, controlled, parallel, examiner-blind clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* You must provide consent to participate by signing this informed consent form.
* Available for the two(2) week study duration.
* You must be at least eighteen(18) years old and not older than seventy(70) years of age.
* You must not smoke.
* You must be in good general health for participation in the study, based on the opinion of the study investigator.
* You must have at least 20 natural permanent teeth.
* Your teeth must meet the scoring entry criteria for dental plaque and gingivitis(gum inflammation) at the discretion of the study examiner.
* You must meet the scoring criteria for gum discomfort, determined using your responses to the survey questionnaire.
* You must have no known history of allergy to personal care/consumer products or their ingredients, relevant to any ingredients in the test products as determined by the study examiner.

Exclusion Criteria:

* Medical condition which requires premedication prior to dental visits/procedures.
* Presence of fix/ removable prosthodontics dentures that may interfere with this study clinical examinations.
* Advanced periodontal disease (gum disease) and/or treatment for periodontal disease (including surgery) within the past twelve months.
* Five (5) or more decayed, untreated dental sites (cavities) and/or any dental condition requiring urgent dental care.

Abnormalities/diseases of the soft or hard oral tissues.

* Orthodontic appliances/bands/lingual bars that interfere with any clinical assessment (plaque scoring)
* Current smokers and/or tobacco users and/or a history of alcohol or drug abuse.
* Use of drugs that can affect salivary flow.
* Use of antibiotics one (1) month prior to study entry and/or during participation in this study.
* Use of any over the counter medications other than analgesics that could interfere with the study at PI discretion.
* Self-reported pregnancy and/or breastfeeding.
* Current Participation in another clinical study or during the month prior to this clinical study entry.
* Known allergies and/or reactions to common dentifrice ingredients.
* Medical condition which prohibits not eating/drinking or chewing gum for four (4) hours prior to your scheduled visits.
* Immunocompromised conditions (AIDS, immunosuppressive drug therapy).
* Infectious disease and/or other blood borne diseases (Hepatitis series, HIV, tuberculosis).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Turesky Modification of the Quigley & Hein Plaque Index | baseline and six months
  Reduction in plaque measurement is served as primary efficacy variable are served. The scoring scheme for the Turesky Modification of the Quigley-Hein dental plaque index is as follows: 0 = no plaque. 1 = separate flecks of plaque at the cervical margin of the tooth. 2 = a thin continuous band of plaque (up to 1 mm) at the cervical margin of the tooth.

SECONDARY OUTCOMES:
questionnaire | six months
  self-reported questionnaires are served as secondary efficacy variable.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Carl Gustav Carus Technische Universität Dresden Department of Periodontology Fetscherstras, Dresden, Germany

IPD SHARING:
Plan to Share IPD: No